CLINICAL TRIAL: NCT06621108
Title: Focus Group Study on the Feeling Tone Mindfulness Course
Status: Not yet recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: 1005240113_Study2b
Record Dates: First submitted 2024-09-16; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Mindfulness; Self-Compassion; Depression; Anxiety; Stress; Well-being
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Focus group session: All participants in this study will take part in a focus group session.
  Interventions: Other: Focus group session

INTERVENTIONS:
Other: Focus group session — Participants will take part in a focus group, which includes sharing their experience of the four-week feeling tone mindfulness course in an online group session. The focus group session will be led by trained moderator, and attended by several other course participants who completed the four-week feeling tone mindfulness course. The session will be audio-recorded as the research team will analyze the qualitative feedback offered by participants.

SUMMARY:
This is an academic research study aiming to explore the acceptability, feasibility, and effectiveness of a four-week feeling tone mindfulness course by gathering qualitative feedback from course participants in a focus group format.

DETAILED DESCRIPTION:
This is a follow-up study of the four-week feeling tone mindfulness course study, exploring the acceptability, feasibility, and effectiveness of the four-week feeling tone mindfulness course by gathering qualitative feedback from course participants in an online (e.g., Zoom), focus group format. A trained moderator will use a semi-structured interview guide with a set of questions to facilitate focus group discussions. Each focus group session will last for about two hours. With the consent from focus group participants, each focus group will be audio-recorded. After participants have completed the focus group, they are eligible to receive HKD100, as a token of thanks to their support and participation to this focus group study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above
* Speak and understand Cantonese as well as written Chinese to a level where the participant can fully take part in the focus group session without the need for translation support
* Have means to access online teleconferencing meeting software (e.g., Zoom), online surveys (to give their informed consent and to schedule a focus group session), online materials, and Short Message Service (SMS) or WhatsApp messenger.
* Participants who have completed the four-week feeling tone mindfulness course

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in this study are adult individuals who have previously completed the four-week feeling tone mindfulness intervention course.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Acceptability and feasibility of the four-week feeling tone mindfulness course, based on an unpublished focus group interview guide at the Department of Psychology, The University of Hong Kong | 4 weeks
  Participants will provide qualitative feedback on the acceptability and feasibility of the four-week feeling tone mindfulness course. Example question will include: "What kept you continue on and complete the course?"
Effectiveness of the four-week feeling tone mindfulness course, based on an unpublished focus group interview guide at the Department of Psychology, The University of Hong Kong | 4 weeks
  Participants will provide qualitative feedback on the effectiveness of the four-week feeling tone mindfulness course. Example question will include: "Now that the course has completed, did it help you attain what you expected?"

CONTACTS AND LOCATIONS:
Overall Officials: Hoi Chun Lok, MSocSc(CP), Principal Investigator — Department of Psychology, The University of Hong Kong
Locations (1):
- Department of Psychology, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No